CLINICAL TRIAL: NCT02382211
Title: A Prospective Observational Trial to Evaluate the Correlation of T-SPOT® Response to CMV Infection and T Cell-mediated Acute Graft Rejection
Brief Title: T-SPOT.CMV and T-SPOT.PRT Diagnostic Assays
Acronym: PROTECT
Status: Completed | Type: Observational
Sponsor: Oxford Immunotec (Industry)
Responsible Party: Sponsor
Other Study IDs: US OI 124
Record Dates: First submitted 2015-02-16; First posted 2015-03-06 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2018-04

CONDITIONS: Infection in Solid Organ Transplant Recipients
Keywords: CMV

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The T-SPOT assay quantifies the number of peripheral blood interferon-γ producing effector T cells [spot forming cells/million peripheral blood mononuclear cells - PBMC)]. The T-SPOT platform technology can be applied to diagnose and monitor any major disease process driven by a T cell response, including a viral disease such as cytomegalovirus (CMV) infection (the T-SPOT.CMV assay) or an allograft rejection (the T-SPOT.PRT assay).

DETAILED DESCRIPTION:
Approximately 600 subjects who meet inclusion/exclusion criteria will be enrolled in the prospective, non-randomized, observational study. Sample size is based on having an adequate overall number of subjects to assess the T-SPOT.PRT endpoint (350) and the T-SPOT.CMV endpoint (250) in the defined populations. Subjects may be enrolled from pre-transplantation to post-transplantation up to completion of antiviral prophylaxis.

Study duration: 37 months; 25 months to enroll all subjects with 12 months (365 days) of patient participation.

Study population:

All subjects enrolled in this study will be men or women, aged 18 years or older and recipients of a first or subsequent renal transplant.

ELIGIBILITY:
Inclusion criteria:

1. Active candidate or recipient of a kidney transplant. Patients enrolled post-transplant must be within 6 months of transplantation and on active CMV anti-viral prophylaxis.
2. Age ≥ 18 years.
3. CMV serology of donor and recipient confirmed prior to enrollment. For seronegative subjects (R-), CMV serostatus should be confirmed within eight weeks prior to transplant by the site local laboratory.
4. Able to provide T-SPOT pre-transplant samples up to a maximum of one month prior to transplant (in the interval between Day -30 and Day 0), or at the time of enrollment if this occurs following transplantation.
5. IRB approved written Informed Consent and privacy language per national regulation (e.g., Health Insurance Portability and Accountability Act for US sites) must be obtained from the subject or legally authorized representative prior to any study related procedures, including screening evaluations and tests.

Exclusion criteria:

1. Anemia prior to transplant that indicates not a candidate for blood draw.
2. On active immunosuppression within two months prior to transplant.
3. Multi-organ transplant (dual-kidney allocation is allowed).
4. Subject has received prior exposure to a CMV vaccine.
5. Subject has undergone or is planning to undergo plasmapheresis.
6. Subject requires desensitization for ABO blood type incompatibility or a positive T or B-cell crossmatch.
7. Subject is known to be HIV positive.
8. Subject is known to have a clinically significant medical or psychiatric condition considered a high risk for participation in an investigational study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active candidate for a kidney transplant. Age equal to or greater than 18 years.
  Male or female.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2015-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Assessment of anti-CMV cell-mediated immunity using the change in T-SPOT counts | Change in T-SPOT counts from baseline to 365 days post transplant.

CONTACTS AND LOCATIONS:
Locations (39):
- United States (35):
  - University of Arizona, Tucson, Arizona
  - University of California, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Transplant Research Institute, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic, Weston, Florida
  - Emory University, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - U Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - U Nebraska, Omaha, Nebraska
  - St Barnabas Medical Center, Livingston, New Jersey
  - Albany Medical Center, Albany, New York
  - Erie County Medical Center, Buffalo, New York
  - ICON School of Medicine at Mt Sinai, New York, New York
  - SUNY, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Case Medical Center, Cleveland, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Legacy Transplant Services, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - Houston Methodist, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Intermoutain Health Care, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
  - Providence Health and Services, Spokane, Washington
- University Health Network, Toronto, Ontario, Canada
- United Kingdom (3):
  - Queen Elizabeth Hospital, Birmingham
  - Guy's Hospital, London
  - Churchill Hospital, Oxford